CLINICAL TRIAL: NCT04370873
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dose MK-5475 in Participants With Pulmonary Hypertension Associated With COPD
Brief Title: Frespaciguat (MK-5475) in Participants With Pulmonary Hypertension Associated With Chronic Obstructive Pulmonary Disease (PH-COPD) (MK-5475-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 5475-006; MK-5475-006 (Other: MSD); 2020-000488-22 (EudraCT Number)
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Part 1 enrolled immediately. Part 2 enrolled following review of Part 1 pharmacokinetic data. A third part was planned but did not enroll because Part 2 yielded sufficient data and Part 3 was optional per protocol.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Frespaciguat (Experimental): Participants receive frespaciguat 360 μg once daily (QD) via inhalation from Days 1-7. Following review of pharmacokinetic (PK) and safety data, a second 7 days of dosing may be initiated. A dose of up to 360 μg up to twice a day may be administered based on PK data in these participants.
  Interventions: Drug: Frespaciguat
- Part 1: Placebo (Placebo Comparator): Participants receive placebo QD via inhalation from Days 1-7.
  Interventions: Drug: Placebo
- Part 2: Frespaciguat (Experimental): Participants receive frespaciguat 32 µg, 100 µg, 195 µg or 380 μg QD via inhalation from Days 1-28.
  Interventions: Drug: Frespaciguat
- Part 2: Placebo (Placebo Comparator): Participants receive placebo QD via inhalation from Days 1-28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frespaciguat — Frespaciguat 32 µg, 100 µg, 195 µg, 360 µg or 380 µg administered as dry powder inhalation according to randomization. Following review of pharmacokinetic (PK) and safety data, a second 7 days of dosing may be initiated. A dose of up to 360 μg up to twice a day may be administered based on PK data. Dosage may be adjusted downwards in Part 2, if indicated by PK results in Part 1.
  Other Names: MK-5475
  Arms: Part 1: Frespaciguat; Part 2: Frespaciguat
Drug: Placebo — Placebo administered as dry powder inhalation according to randomization
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The primary objectives of this study are to assess the safety/tolerability and efficacy (by evaluating changes in pulmonary vascular resistance [PVR] and pulmonary blood volume [PBV]) of frespaciguat in participants with pulmonary hypertension associated with chronic obstructive pulmonary disease (PH-COPD). The primary hypothesis is that 28 days of frespaciguat treatment is superior to placebo treatment in reduction of PVR.

DETAILED DESCRIPTION:
Part 1 of this study will assess safety, tolerability, and PK of frespaciguat compared to placebo. Part 2 will assess safety, tolerability, PK, and changes in PVR and PBV of frespaciguat compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, from 40 to 80 years of age inclusive at the time of signing informed consent.
* Be judged to have no untreated, clinically significant health issue from other comorbidities based on medical history, physical examination, vital signs and electrocardiograms performed at the screening visit(s)
* Be judged to have no untreated, clinically significant health issue from other comorbidities based on laboratory safety tests performed at the screening visit(s)
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 14 days, corresponding to time needed to eliminate study intervention(s) (eg, 5 terminal half-lives) plus an additional 90 days (a spermatogenesis cycle) after the last dose of study intervention. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or agrees to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: She is a woman of nonchildbearing potential (WONCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis)
* Have been diagnosed with mild to severe Chronic Obstructive Pulmonary Disease (COPD) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) diagnostic criteria (postbronchodilator forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC) ratio < 0.7)
* Has Modified Medical Research Council (MMRC) Dyspnea Score in the range of 1 through 3 at screening
* Be deemed clinically stable by the investigator
* Be or have suspected Pulmonary Hypertension Group 3 in particular: COPD
* Have a history of right heart catheterization (RHC) within 3 years of starting study medication demonstrating mean pulmonary artery pressure (mPAP) ≥ 25mmHg and pulmonary vascular resistance (PVR) ≥ 3.75 Woods units or 300 dynes/sec/cm or have an echocardiogram performed by the investigator (or appropriate designee) at screening or within 1 year of screening demonstrating pulmonary artery systolic pressure ≥ 38 mmHg (Part 1 only) or ≥ 50 mmHg (Part 2 only) in conjunction with one or more of the following: tricuspid regurgitation velocity >3 m/s or significant right heart enlargement and or reduced right heart function

Exclusion Criteria:

* Has pulmonary hypertension subtypes including the following according to Nice 2013 Clinical classification. This includes Group 1 Pulmonary arterial hypertension (PAH): Idiopathic PAH, Heritable PAH including Bone morphogenetic protein receptor type II (BMPR2), Activin A receptor type II-like kinase-1 (ALK1), endoglin, Sterile alpha motif domain-containing protein 9 (SMAD9), caveolin 1 (CAV1), potassium two-pore-domain channel subfamily K member 3 (KCNK3) and unknown, Drug and toxin-induced PAH, PAH associated with Connective tissue disease, HIV infection, Portal hypertension, Congenital heart disease (unrepaired and not requiring repair or repaired simple cardiac defects at least 1year status post corrective surgery, with no clinically significant residual shunt), Schistosomiasis, Chronic hemolytic anemia, Persistent pulmonary hypertension of the newborn (PPHN), and Pulmonary veno-occlusive disease (PVOD) and or pulmonary capillary hemangiomatosis (PCH); Group 2 Pulmonary hypertension owing to left heart diseases including Left ventricular Systolic dysfunction, Left ventricular Diastolic dysfunction, Valvular disease, Congenital/acquired left heart inflow/outflow tract obstruction and congenital cardiomyopathies; Group 3 Pulmonary hypertension owing to lung diseases or hypoxia not associated with COPD including Interstitial lung disease, Other pulmonary diseases with mixed restrictive and obstructive pattern, Sleep-disordered breathing (mild obstructive sleep apnea (OSA) may be permitted with sponsor consultation), Alveolar hypoventilation disorders. Chronic exposure to high altitude, Developmental abnormalities; Group 4 Pulmonary hypertension defined as Chronic thromboembolic pulmonary hypertension [CTEPH]); and Group 5 Pulmonary Hypertension with unclear multifactorial mechanisms including Hematologic disorders: chronic hemolytic anemia, myeloproliferative disorders, Splenectomy, Systemic disorders: sarcoidosis, pulmonary Langerhans cell histiocytosis, lymphangioleimyomatosis, neurofibromatosis, vasculitis, Metabolic disorders: glycogen storage disease, Gaucher disease, thyroid disorders, and Others: tumoral obstruction, fibrosing mediastinitis, chronic renal failure, segmental pulmonary hypertension.
* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic (not including chronic stable Hep B and C), immunological, renal, respiratory (not including PH-COPD), genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems at the time of pre-study (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator
* Has a history of cancer (malignancy) except adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, in the opinion of the investigator and with agreement of the Sponsor
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or non-prescription drugs or food
* Is positive for hepatitis B surface antigen (HBsAg) [acute infection] or HIV (participants with positive HBsAG that demonstrate low viral load (chronic stable infection) are permitted.
* Part 2 only: Has known sensitivity to iodine or iodine containing products
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has persistent or permanent atrial fibrillation with uncontrolled ventricular rate (participants with paroxysmal atrial fibrillation or controlled atrial fibrillation with no clinically significant arrhythmia may be allowed per the judgement of the investigator)
* Has history of combined pulmonary fibrosis and emphysema (CPFE) or severe bullous emphysema. If no history, a confirmed negative high-resolution computerized tomography scan (HRCT) for these conditions needs to have been performed within last 2 ears.
* Has an active respiratory infection (common cold, influenza, pneumonia, acute bronchitis) with lung function values (FEV1 and/or FEV1/FVC ratio) that do not meet eligibility range
* Has a physical limitation that will inhibit the participant to effectively perform low intensity exercise testing (e.g. severe arthritis of the hip or knee)
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the poststudy visit. There may be certain medications that are permitted
* Is currently on monotherapy calcium channel blockers as a specific treatment for pulmonary hypertension
* Is currently taking nitrates, inhaled prostacyclin, immediate or extended release diltiazem, phosphodiesterase 5 (PDE5) inhibitors or soluble guanylate cyclase (sGC) or activators for the treatment of pulmonary hypertension. Participants previously using medications to treat pulmonary arterial hypertension may be enrolled provided they have been off therapy for at least 2 weeks prior to the start of the screening period
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit. The window will be derived from the date of the last visit in the previous study
* Has FEV1 < 30% predicted based on Pulmonary Function Tests (PFTs) at screening
* Part 2 only: Does not meet RHC criteria at baseline
* Participant has an estimated creatinine clearance of < 60 mL/min based on the Cockcroft Gault equation at screening
* Suffers from claustrophobia and is unable to undergo a computerized tomography (CT) scan
* Has participated in a positron emission tomography (PET) research study or other research study involving administration of a radioactive substance or ionizing radiation within 12 months prior to the screening visit or has undergone or plans to have extensive radiological examination within the period with a radiation burden over 10 millisievert (mSv)
* Does not agree to follow the smoking restrictions as defined by the clinical research unit (CRU)
* Consumes greater than 3 glasses of alcoholic beverages
* Consumes excessive amounts, defined as greater than 6 servings of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months. Participants must have a negative urine drug screen (UDS) prior to randomization

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- United States (6):
  - Lexington VA- Health Care System ( Site 0034), Lexington, Kentucky
  - Johns Hopkins - University ( Site 0003), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 0005), Boston, Massachusetts
  - Brigham & Women's Hospital ( Site 0001), Boston, Massachusetts
  - University of Rochester Medical Center ( Site 0012), Rochester, New York
  - Medical Universtiy of South Carolina ( Site 0011), Charleston, South Carolina
- Israel (2):
  - Rambam Medical Center ( Site 0037), Haifa
  - Rabin Medical Center ( Site 0035), Petah Tikva
- Republican Clinical Hospital of Moldova ( Site 0013), Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Bajwa EK, Cislak D, Kumar A, Li D, Messina EJ, Reynders T, Denef JF, Corcea V, Buch KP, Lai E, Stoch SA. Phase 1 Study of MK-5475, an Inhaled Soluble Guanylate Cyclase Stimulator, in Participants with Pulmonary Hypertension Associated with Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2024 May 23;19:1105-1121. doi: 10.2147/COPD.S454905. eCollection 2024. PMID 38803412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with pulmonary hypertension (PH) associated with chronic obstructive pulmonary disease (COPD) were recruited to evaluate safety, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple doses of MK-5475.
Pre-assignment Details: There were three planned parts in the study. Participants in part 1 received MK-5475 360 μg. Participants in part 2 received MK-5475 380 μg. Part 3 was not performed because, as allowed by the protocol, it was decided that sufficient data had already been obtained. One participant in Part 1 also participated in Part 2. That participant is counted only in Part 1 for the participant flow.
Groups:
- Part 1: MK-5475 360 μg: Participants received MK-5475 360 μg once daily (QD) via inhalation from Days 1-7.
- Part 1: Placebo: Participants received placebo QD via inhalation from Days 1-7.
- Part 2: MK-5475 380 μg: Participants received MK-5475 380 μg QD via inhalation from Days 1-28.
- Part 2: Placebo: Participants received placebo QD via inhalation from Days 1-28.
Period: Part 1: 7-day Dosing
Arm/Group | Part 1: MK-5475 360 μg | Part 1: Placebo | Part 2: MK-5475 380 μg | Part 2: Placebo
Started | 6 | 3 | 0 | 0
Completed | 6 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2: 28-day Dosing
Arm/Group | Part 1: MK-5475 360 μg | Part 1: Placebo | Part 2: MK-5475 380 μg | Part 2: Placebo
Started | 0 | 0 | 8 | 5
Completed | 0 | 0 | 8 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant in Part 1 also participated in Part 2. That participant is counted only in Part 1 for baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-5475 360 μg | Part 1: Placebo | Part 2: MK-5475 380 μg | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 3 | 8 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (12.7) | 62.3 (8.7) | 69.4 (4.8) | 66.6 (5.6) | 65.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 3
  Male | 5 | 1 | 8 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 8 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 3 | 8 | 5 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Pulmonary Vascular Resistance (PVR): Part 2 [Mean (Standard Deviation); unit: dynes*s*cm^-5] — PVR was calculated in participants at baseline in participants who underwent right heart catheterization (RHC) via thermodilution. Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and complied with the protocol without major protocol deviations.
  dynes*s*cm^-5
    number analyzed (Participants) | 0 | 0 | 8 | 4 | 12
    (all) |  |  | 409.52 (166.47) | 394.32 (141.18) | 404.46 (152.08)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE was assessed.
Time Frame: Up to approximately 139 days
Population: All participants who received ≥1 dose of investigational treatment were analyzed according to treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: MK-5475 360 μg | Part 1: Placebo | Part 2: MK-5475 380 μg | Part 2: Placebo
Number analyzed (Participants) | 6 | 3 | 9 | 5
Percentage of Participants | 33.3 | 33.3 | 33.3 | 80.0

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to approximately 32 days
Population: All participants who received ≥1 dose of investigational treatment were analyzed according to treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: MK-5475 360 μg | Part 1: Placebo | Part 2: MK-5475 380 μg | Part 2: Placebo
Number analyzed (Participants) | 6 | 3 | 9 | 5
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Percentage Change From Baseline to Day 28 in Pulmonary Vascular Resistance (PVR): Part 2
Description: PVR was calculated in participants after MK-5475 dosing at baseline and Day 28. Based on the variables obtained by right heart catheterization (RHC), the fold change from baseline individual PVR was calculated. The difference from baseline was assessed on the log scale and then back-transformed for reporting (percent change from baseline). Per protocol, this outcome measure was only assessed during the Part 2 and was not assessed during part 1.
Time Frame: Baseline (between Day -5 and Day -1) and Day 28
Population: All Part 2 participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available data at baseline and Day 28.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Part 2: MK-5475 380 μg | Part 2: Placebo
Number analyzed (Participants) | 8 | 4
Percentage change | -21.23 (16.98) | -5.39 (49.21)

4. Secondary Outcome: Plasma Area Under the Concentration Time-Curve From 0 to Infinity (AUC0-inf) of MK-5475: Part 1
Description: Blood samples were taken predose and at specified times postdose to determine the AUC0-inf of MK-5475. Plasma AUC0-inf was defined as the area under the concentration vs. time curve for MK-5475 from 0 to infinite hours.
Time Frame: Day 1: Predose, 5 minutes, 15 minutes, 0.5, 1, 2, 3, 4 and 8 hours postdose, Day 7: Predose, 5 minutes, 15 minutes, 0.5, 1, 2, 3, 4, 8 and 24 hours postdose
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of AUC0-inf. Per protocol, AUC0-inf was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
hr*nM
  Day 1 | 3.32 (68.9)
  Day 7 | 4.03 (90.2)

5. Secondary Outcome: Plasma Area Under the Concentration Time-Curve From 0 to 24 Hours (AUC0-24) of MK-5475: Part 1
Description: Blood samples were taken predose and at specified times postdose on Day 7 to determine the AUC0-24 of MK-5475. AUC0-24 values for Day 1 correspond to extrapolated values since collection on Day 1 stopped at 8 hours.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of AUC0-24. Per protocol, AUC0-24 was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
hr*nM
  Day 1 | 3.31 (68.7)
  Day 7 | 4.22 (83.5)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MK-5475: Part 1
Description: Plasma concentration of MK-5475 was quantified for each arm to determine Cmax.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of Cmax. Per protocol, Cmax was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
nM
  Day 1 | 0.830 (50.8)
  Day 7 | 0.970 (59.1)

7. Secondary Outcome: Plasma Concentration 24 Hours Postdose (C24) of MK-5475: Part 1
Description: Blood samples were taken to determine the C24 of MK-5475. Data are reported as Mean with Standard Deviation. Concentration values below the lower limit of quantification were treated as having a value of 0.
Time Frame: 24 hours postdose on Day 7
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of C24. Per protocol, C24 was calculated for the participants who had concentration.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
nM | 0.02 (0.3)

8. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-5475: Part 1
Description: Blood samples were taken at predose and at specified time points postdose to determine the Tmax of MK-5475. Tmax was defined as the time to maximum concentration of MK-5475.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of Tmax. Per protocol, Tmax was calculated for the participants who had concentration values.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
Hours
  Day 1 | 1.00 [1.00 to 2.00]
  Day 7 | 1.00 [1.00 to 2.00]

9. Secondary Outcome: Plasma Apparent Terminal Half-Life (t½) of MK-5475: Part 1
Description: Blood samples were taken at predose and at specified time points postdose to determine the t½ of MK-5475.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of t½. Per protocol, t½ was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
Hours
  Day 1 | 2.13 (18.5)
  Day 7 | 2.81 (48.4)

10. Secondary Outcome: Cmax Accumulation Ratio of MK-5475: Part 1
Description: Blood samples were taken predose and at specified times postdose to determine the Cmax accumulation ratio of MK-5475. Accumulation ratio is the ratio of the Day 7 Cmax to the Day 1 Cmax.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of Cmax accumulation ratio. Per protocol, Cmax accumulation ratio was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
Ratio | 1.17 (28.8)

11. Secondary Outcome: AUC0-24 Accumulation Ratio of MK-5475: Part 1
Description: Blood samples were taken predose and at specified times postdose to determine the AUC0-24 accumulation ratio of MK-5475. Accumulation ratio is the ratio of the Day 7 AUC0-24 to the Day 1 AUC0-24.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of AUC0-24 accumulation ratio. Per protocol, AUC0-24 accumulation ratio was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
Ratio | 1.27 (30.1)

12. Secondary Outcome: AUC0-inf Accumulation Ratio of MK-5475: Part 1
Description: Blood samples were taken predose and at specified times postdose on Days 1-7 to determine the AUC0-inf accumulation ratio of MK-5475. Accumulation ratio is the ratio of the Day 7 AUC0-inf to the Day 1 AUC0-inf.
Time Frame: as for outcome 4
Population: The analysis population consisted of all participants in part 1 who received at least one dose of MK-5475 360 μg and who contributed blood samples for analysis of AUC0-inf accumulation ratio. Per protocol, AUC0-inf accumulation ratio was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: MK-5475 360 μg
Number analyzed (Participants) | 6
Ratio | 1.21 (31.1)

13. Secondary Outcome: AUC0-inf of MK-5475: Part 2
Description: Blood samples were taken pre-dose and at specified times post-dose to determine the AUC0-inf of MK-5475. Concentrations for samples collected pre-RHC in a time window of 6-8 hours postdose on Day 28 were used to derive PK parameter values on Day 28. A nominal elapsed time of 6.01 hours postdose was used in the calculation.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of AUC0-inf. Per protocol, AUC0-inf was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
hr*nM
  Day 1 | NA (NA) — NA= AUC0-inf could not be calculated due to insufficient data.
  Day 28 | 1.98 (105.9)

14. Secondary Outcome: AUC0-24 of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose on Day 28 to determine the AUC0-24 of MK-5475. Concentrations for samples collected pre-RHC in a time window of 6-8 hours postdose on Day 28 were used to derive PK parameter values on Day 28. A nominal elapsed time of 6.01 hours postdose was used in the calculation. AUC0-24 was calculated using extrapolated concentration at 24 hours postdose.
Time Frame: Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of AUC0-24. Per protocol, AUC0-24 was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
hr*nM
  Day 1 | NA (NA) — NA= AUC0-24 could not be calculated due to insufficient data.
  Day 28 | 1.97 (105.7)

15. Secondary Outcome: Cmax of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose to determine the Cmax of MK-5475.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of Cmax. Per protocol, Cmax was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
nM
  Day 1 | 0.348 (48.4)
  Day 28 | 0.397 (71.4)

16. Secondary Outcome: Plasma Concentration 24 Hours Postdose (C24) of MK-5475: Part 2
Description: Blood samples were taken to determine the C24 of MK-5475. Data are reported as Mean with Coefficient of Variation, but due to data entry limitations the table below labels them as Geometric Mean and Geometric Coefficient of Variation. Concentration values below the lower limit of quantification were treated as having a value of 0.
Time Frame: 24 hours postdose on Day 7
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of C24. Per protocol, 24 hours samples were not collected. Therefore, no participants were analyzed.
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 0

17. Secondary Outcome: Tmax of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose to determine the Tmax of MK-5475.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of Tmax. Per protocol, Tmax was calculated for the participants who had concentration values.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
Hours
  Day 1 | 1.50 [1.00 to 2.00]
  Day 28 | 1.50 [1.00 to 2.00]

18. Secondary Outcome: t½ of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose to determine the t½ of MK-5475.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of t½. Per protocol, t½ was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
Hours
  Day 1 | NA (NA) — NA= t½ could not be calculated due to insufficient data.
  Day 28 | 2.06 (62.4)

19. Secondary Outcome: AUC0-3 Accumulation Ratio of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose on to determine the AUC0-3 accumulation ratio of MK-5475. Accumulation ratio is the ratio of the Day 7 AUC0-3 to the Day 1 AUC0-3.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants who received at least 1 treatment and who contributed blood samples for analysis of accumulation. Per protocol, accumulation was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
Ratio | 1.11 (53.8)

20. Secondary Outcome: Cmax Accumulation Ratio of MK-5475: Part 2
Description: Blood samples were taken predose and at specified times postdose to determine the Cmax accumulation ratio of MK-5475. Cmax accumulation ratio is the ratio of the Day 7 Cmax to the Day 1 Cmax.
Time Frame: Day 1: Predose, 0.5, 1, 2 and 3 hours postdose, Day 15: 1 hour postdose, Day 28: Predose, 0.5, 1, 2 and 3 hours postdose
Population: The analysis population consisted of all participants in part 2 who received at least one dose of MK-5475 380 μg and who contributed blood samples for analysis of Cmax accumulation ratio. Per protocol, Cmax accumulation ratio was calculated for the participants who had concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: MK-5475 380 μg
Number analyzed (Participants) | 8
Ratio | 1.14 (51.6)

21. Secondary Outcome: Percent Change From Baseline in Pulmonary Blood Volume (PBV) at Day 28: Part 2
Description: Participants underwent a series of computed tomography (CT) scans with an intravenous (IV) iodinated contrast agent to facilitate assessment of PBV at baseline and at several times points after MK-5475 dosing. Percentage change from baseline (CFB) in PBV was calculated and reported for each dose group that underwent FRI in Part 2. As pre-specified, central tendency for PBV percentage CFB was provided as numerical values rounded to whole numbers. Per protocol, this outcome measure was only assessed during the Part 2 FRI Period for each panel and was not assessed during part 1 and part 3.
Time Frame: Baseline (between Day -5 and Day -1) and Day 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2: MK-5475 380 μg | Part 2: Placebo
Number analyzed (Participants) | 9 | 5
Percentage Change | -0.3 (4.7) | -2.8 (10.6)

ADVERSE EVENTS:
Time Frame: Up to approximately 139 days
Description: All-cause mortality includes all randomized participants and adverse events include all participants who received at least one dose of study treatment.
Groups:
- MK-5475 360 µg (Part 1): Participants received MK-5475 360 μg once daily (QD) via inhalation from Days 1-7.
- Placebo (Part 1): Participants received placebo QD via inhalation from Days 1-7.
- MK-5475 380 µg (Part 2): Participants received MK-5475 380 μg QD via inhalation from Days 1-28.
- Placebo (Part 2): Participants received placebo QD via inhalation from Days 1-28.
Arm/Group | MK-5475 360 µg (Part 1) | Placebo (Part 1) | MK-5475 380 µg (Part 2) | Placebo (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 1/9 | 1/5
Other Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 2/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5475 360 µg (Part 1) (N=6) | Placebo (Part 1) (N=3) | MK-5475 380 µg (Part 2) (N=9) | Placebo (Part 2) (N=5)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5475 360 µg (Part 1) (N=6) | Placebo (Part 1) (N=3) | MK-5475 380 µg (Part 2) (N=9) | Placebo (Part 2) (N=5)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT04370873/Prot_SAP_000.pdf